CLINICAL TRIAL: NCT03261765
Title: Effect of Multiple Repeat Cesarean Sections on Intra-abdominal Adhesions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, principal investigator, Assiut University
Other Study IDs: CSIAA
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Cesarean Section Complications

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Multiple repeat cesarean (four or more)
  Interventions: Other: Assessment of adhesions
- Fewer repeat cesarean (two-three)
  Interventions: Other: Assessment of adhesions

INTERVENTIONS:
Other: Assessment of adhesions — Modified Nair scoring system

SUMMARY:
The rate of cesarean section deliveries has increased dramatically worldwide in the last decades. While the cesarean birth rate was 4.5% in the USA in 1965, it was 31.8% according to 2007 data and is thought to be over 50% at present. The reasons for this include advanced age of primigravida, a wide range of indications, patient requests, the frequency of women with previous cesareans, women's rejections to offers of sterilization, and the common usage of assisted reproductive techniques

ELIGIBILITY:
Inclusion Criteria:

1. Women with at least previous one cesarean section.
2. Women accepted to participate in the study.

Exclusion Criteria:

1. Previous abdominopelvic surgery other than cesarean section.
2. History of Pelvic inflammatory disease.
3. Women refuse to participate in the study.
4. Intrauterine fetal death

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All women with repeated cesarean section
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Rate of abdominal adhesions | 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No